CLINICAL TRIAL: NCT00244465
Title: Post Marketing Non-interventional Surveillance Pharmacoepidemiology Study (PMSS) to Evaluate Long-term Safety, Tolerability and Compliance in Administration of Xyrem® (Sodium Oxybate) Oral Solution in Patients Who Receive Treatment With This Medication in Regular Clinical Practice.
Brief Title: Observational Study to Evaluate Risks of Side Effects, Drug Abuse and Dependence in Patients Who Received Xyrem ® on Prescription
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: C00302
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; Cataplexy; Oxybate; Xyrem; Misuse; Safety
MeSH Terms: conditions — Narcolepsy; Cataplexy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients will be followed up for max 18 months. Information on the Adverse Events and potential misuse or abuse of Xyrem ® will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Xyrem ® on prescription

Exclusion Criteria:

* No limitations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients being treated with Xyrem®.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2006-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of risk for development adverse events, withdrawal syndrome and potential for dependence, abuse, overdose and misuse of Xyrem®. Obtaining information about adherence to Xyrem® prescribing information regarding indication and dosage. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (41):
- Austria (2):
  - 9, Graz
  - 5, Innsbruck
- Belgium (6):
  - 12, Antwerp
  - 28, Bruges
  - 13, Brussels
  - 34, Ghent
  - 35, Leuven
  - 10, Liège
- 16, Prague, Czechia
- Germany (10):
  - 24, Berlin
  - 25, Berlin
  - 22, Bremen
  - 19, Hofheim/Taunus
  - 42, Katzenelnbogen
  - 23, Münster
  - 20, Regensburg
  - 1, Schwalmstadt
  - 31, Ulm
  - 21, Westerstede
- 4, Dublin, Ireland
- 18, Bologna, Italy
- Spain (14):
  - 40, Barakaldo
  - 11, Barcelona
  - 7, Barcelona
  - 17, Castellon
  - 36, Donostia / San Sebastian
  - 32, Granada
  - 15, Madrid
  - 29, Madrid
  - 39, Palma de Mallorca
  - 14, Seville
  - 37, Seville
  - 38, Vigo
  - 30, Vitoria-Gasteiz
  - 43, Vitoria-Gasteiz
- Switzerland (3):
  - 41, Barmelweid
  - 33, Bern
  - 6, Zurich
- United Kingdom (3):
  - 2, Cambridge
  - 26, Essex
  - 27, Leicester

REFERENCES:
- [Derived] Mayer G, Plazzi G, Iranzo A, Ortega-Albas J, Quinnell T, Pesch H, Serralheiro P, Schlit AF, Wuiame D, Bentz JWG. Long-term compliance, safety, and tolerability of sodium oxybate treatment in patients with narcolepsy type 1: a postauthorization, noninterventional surveillance study. Sleep. 2018 Sep 1;41(9). doi: 10.1093/sleep/zsy128. PMID 29986085